CLINICAL TRIAL: NCT05410067
Title: Effects of Cervicothoracic Junction Mobilization Versus Eccentric Muscle Energy Technique in the Treatment of Mechanical Cervical Pain
Brief Title: Cervicothoracic Junction Mobilization Versus Eccentric Muscle Energy Technique in Mechanical Cervical Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ayesha Sadiq
Record Dates: First submitted 2022-06-04; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervicothoracic Junction Mobilization Technique (Experimental): It is a part of manual therapy technique. Maitland mobilization to the C7- T1 level, according to their primary movement restriction (for flexion-extension restriction- central PA glide, for rotation restrictions unilateral PA glide) is given.For central PA glide, a central pressure angled towards the participant's head was given with overlapping thumbs of the therapist placed on the spinous process of C7.
  Dosage:
  Glide would be given according to the nature, intensity and severity of the patient's pain. 30 sec bouts with 3 sets & 2 reps. Total 2-3 min duration. 2 sessions per week for 3 weeks.
  Interventions: Other: Cervicothoracic Junction Mobilization Technique
- Eccentric Muscle Energy Technique (Experimental): Eccentric muscle energy technique would be applied to the patient's cervical spine. The cervical spine would be brought to the barrier of motion in each plane i.e. flexion/extension, lateral bending and rotation. Then patient would be asked to push their heads into the direction opposite that of the barrier.
  Dosage:
  The therapist provided isometric resistance for 3- 5 seconds, after which the subjects relaxed their muscles completely and the therapist applied stretch. This is applied for generalized cervical movements in each plane like Flexion, Extension, Side Bending
  & Rotation. 3-5 repetitions with 2-3 sets were performed. Total duration: 3-5 min 2 sessions per week for 3 weeks.
  Interventions: Other: Eccentric Muscle Energy Technique

INTERVENTIONS:
Other: Cervicothoracic Junction Mobilization Technique — It is a part of manual therapy technique. Patient would be in prone position with his forehead in the palm of the therapist. Maitland mobilization to the C7- T1 level, according to their primary movement restriction (for flexion-extension restriction- central PA glide, for rotation restrictions unilateral PA glide) is given. For central PA glide, a central pressure angled towards the participant's head was given with overlapping thumbs of the therapist placed on the spinous process of C7. The therapist's thumbs were placed on the posterior surface of the articular process to be mobilized (C7 on the side of restriction), and anteriorly directed oscillatory pressure was applied for unilateral PA mobilization.
  Arms: Cervicothoracic Junction Mobilization Technique
Other: Eccentric Muscle Energy Technique — Eccentric muscle energy technique would be applied to the patient's cervical spine. The cervical spine would be brought to the barrier of motion in each plane i.e. flexion/extension, lateral bending and rotation. Then patient would be asked to push their heads into the direction opposite that of the barrier.
  Arms: Eccentric Muscle Energy Technique

SUMMARY:
1. To compare the effectiveness of the cervicothoracic junction mobilization and eccentric muscle energy technique on mechanical cervical pain.
2. To compare the effectiveness of the cervicothoracic junction mobilization and eccentric muscle energy technique on cervical disability.
3. To compare the effectiveness of the cervicothoracic junction mobilization and eccentric muscle energy technique on cervical ROM.

ELIGIBILITY:
Inclusion Criteria:

* Participants falling in this category would be recruited into the study.

  1. Females
  2. Age between 18-45 years.
  3. Diagnosed with mechanical cervical pain.

Exclusion Criteria:

* Participant failing to fall in this category would be excluded of the study.

  1. Pregnant Females
  2. Any previous history of trauma or surgery
  3. Diagnosed with mechanical cervical pain due to disc herniation, radiculopathy or any other cervical malignancy.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Diagnosed with mechanical cervical pain.
Enrollment: 36 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 3 Weeks
  A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms. It is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom, pain, health) orientated from the left (worst) to the right (best). Test-retest reliability has been shown to be good, but higher among literate (r= 0.94)
Neck Disability Index (NDI) | 3 Weeks
  This questionnaire has been designed to give us information as to how your neck pain has affected your ability to manage in everyday life. Patient-completed, condition-specific, functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation. Each section is scored on a 0 to 5 rating scale, in which zero means "no pain" and 5 means "Worst imaginable pain". It has highest score of 50.
Cervical Goniometer | 3 Weeks
  A goniometer is an instrument which measures the available range of motion atjoint. Goniometer have different types; the most use is the universal standard goniometer, which is either made with plastic or metal tool. It consists of a stationary arm, a movable arm and a fulcrum.

CONTACTS AND LOCATIONS:
Overall Officials: Waqar Ahmad Awan, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah international University, Islamabad, ICT, Pakistan

IPD SHARING:
Plan to Share IPD: No